CLINICAL TRIAL: NCT00472212
Title: Correction of Hyperopia in Children Study
Brief Title: Correction of Farsightedness in Children Study
Acronym: CHICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: American Academy of Optometry (Other); Transitions (Industry); Ohio Lions Eye Research Foundation (Other); College of Optometrists in Vision Development (Other); SUNY Research Foundation (Other)
Responsible Party: Principal Investigator, Marjean Kulp, Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2001H0401
Record Dates: First submitted 2007-05-09; First posted 2007-05-11 (Estimated); Results first posted 2022-08-29 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Hyperopia; Farsightedness
MeSH Terms: conditions — Hyperopia | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spectacles (Experimental): Spectacles with hyperopic lenses
  Interventions: Device: Spectacles
- Control (Placebo Comparator): Spectacles with placebo lenses
  Interventions: Device: Control

INTERVENTIONS:
Device: Spectacles — Hyperopic spectacle lenses
  Arms: Spectacles
Device: Control — Plano (no power, control) spectacle lenses
  Arms: Control

SUMMARY:
The Correction of Hyperopia In Children Study (CHICS) is a placebo-controlled, randomized, masked investigation of the effect of spectacle correction for moderate amounts of hyperopia on visual function, attention, and reading skills in children.

DETAILED DESCRIPTION:
Hyperopia (farsightedness) has been reported to be associated with reduced visual perceptual and reading abilities. However, there is controversy regarding whether or not to prescribe for low to moderate amounts of hyperopia. The Correction of Hyperopia In Children Study (CHICS) is a placebo-controlled, randomized, masked investigation of the effect of spectacle correction for moderate amounts of hyperopia on visual function, attention, and reading skills in children.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-11 years;
* At least +1.00D Hyperopia (farsightedness);
* < +4.00D Hyperopia;
* < 1.00D Astigmatism;
* < 1.00D Anisometropia (difference between the two eyes);
* Willing to be randomized;
* Best corrected visual acuity of 20/25 or better in each eye;
* Willing to wear eyeglasses full-time;
* Willing to return for follow-up visits

Exclusion Criteria:

* Previous wear of glasses or contacts for farsightedness/hyperopia;
* Eye disease that affects visual function;
* Amblyopia (lazy eye);
* Strabismus (eye turn);
* History of strabismus surgery;
* Chronic use of any of the following medications:

  * Antianxiety agents (Librium, Valium)
  * Antiarrythmic agents (Cifenline, Cibenzoline)
  * Anticholinergics (Motion sickness patch - scopolamine)
  * Bladder spasmolytic (Propiverine)
  * Chloroquine
  * Phenothiazines (Compazine, Mellaril, Thorazine)
  * Tricyclic antidepressants (Elavil, Nortriptyline, Tofranil)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2003-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marjean Kulp, OD, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - Illinois College of Optometry/Illinois Eye Institute, Chicago, Illinois
  - SUNY College of Optometry/University Optometric Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Southern College of Optometry, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Glasses With Hyperopic Lenses: Spectacles with hyperopic lenses
  Spectacles: Hyperopic spectacle lenses
Period: Overall Study
Arm/Group | Glasses With Hyperopic Lenses | Control
Started | 31 | 27
Completed | 25 | 23
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glasses With Hyperopic Lenses | Control | Total
Number analyzed (Participants) | 31 | 27 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.58 (1.78) | 7.41 (1.47) | 7.5 (1.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 14 | 14 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: One subject with race /ethnicity not reported
  Participants
    African American: number analyzed (Participants) | 30 | 27 | 57
    African American | 18 | 17 | 35
    White: number analyzed (Participants) | 30 | 27 | 57
    White | 8 | 9 | 17
    Hispanic: number analyzed (Participants) | 30 | 27 | 57
    Hispanic | 4 | 1 | 5
Kaufman Test of Educational Achievement (K-TEA) Reading Comprehension Score [Mean (Standard Deviation); unit: units on a scale (standard score)] — Baseline vision and baseline educational testing completed at separate visits. The Kaufman Test of Educational Achievement (K-TEA) was used to measure change in reading skills (decoding and reading comprehension). The K-TEA is a well-established, individually administered, standardized test for assessment of achievement in reading, with a mean standard score of 100 and standard deviation of 15. Higher values represent better performance. Population: Test results not available for two subjects.
  units on a scale (standard score)
    number analyzed (Participants) | 29 | 27 | 56
    (all) | 95.17 (13.47) | 97.07 (13.38) | 96.09 (13.34)
Cognitive Assessment System (CAS) Attention Score [Mean (Standard Deviation); unit: units on a scale (standard score)] — Baseline vision and baseline educational testing completed at separate visits. The Cognitive Assessment System (CAS) is a well-researched, norm-referenced measure of cognitive ability. Standard scores are normed to a mean of 100 and a standard deviation of 15 for each battery. The CAS attention battery (Expressive Attention, Number Detection, and Receptive Attention) require the participant to selectively attend to a particular stimulus and inhibit attending to competing stimuli. Higher values represent better performance. Population: Test results not available for 2 subjects.
  units on a scale (standard score)
    number analyzed (Participants) | 29 | 27 | 56
    (all) | 97.83 (17.09) | 101.96 (19.52) | 99.82 (18.25)
Accommodative Response by monocular estimation method (MEM) [Mean (Standard Deviation); unit: diopters] — Accommodative response, Right eye. Baseline vision and educational testing completed on separate dates. This technique is used to measure the accuracy of focusing (accommodative response) while the subject views a near target. Lower (positive) values represent better accuracy of focusing.
  diopters | 0.71 (0.42) | 0.67 (0.45) | 0.69 (0.43)

OUTCOME MEASURES:

1. Primary Outcome: Change in Kaufman Test of Educational Achievement (K-TEA) Reading Comprehension Score as Measured From Baseline to After 6 Weeks of Assigned Treatment (Hyperopic or Control Correction)
Description: The Kaufman Test of Educational Achievement (K-TEA) was used to measure change in reading skill (reading comprehension). The K-TEA is a well-established, individually administered, standardized test for assessment of achievement in reading, with a mean standard score of 100 and standard deviation of 15. Higher values represent better performance.
Time Frame: 6 week outcome exam
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Glasses With Hyperopic Lenses: Glasses with hyperopic lenses (Correction)
- Control: Glasses with placebo lenses
  Control: Glasses with plano (no power, control) spectacle lenses
Arm/Group | Glasses With Hyperopic Lenses | Control
Number analyzed (Participants) | 24 | 23
score on a scale | -2.92 [-7.9 to 2.1] | 0.088 [-5.0 to 5.2]

2. Secondary Outcome: Change in Cognitive Assessment System (CAS) Attention Scores as Measured From Baseline to After 6 Weeks of Assigned Treatment (Hyperopic or Control Correction)
Description: Individually administered battery designed to measure cognitive processing abilities. CAS is based on PASS (Planning, Attention, Simultaneous, and Successive), a well-researched cognitive/neuropsychological theory.
  A higher score indicates a better outcome.
Time Frame: 6 week outcome exam
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Glasses With Hyperopic Lenses | Control
Number analyzed (Participants) | 24 | 23
score on a scale | 9.14 [4.8 to 13.5] | 3.46 [-1.0 to 7.9]

3. Secondary Outcome: Change in Accommodative Response From Baseline to After 6 Weeks of Assigned Treatment (Hyperopic or Control Correction)
Description: Accommodative response, Right eye. This is a measure the accuracy of focusing (accommodative accuracy or response) while the subject views a near target. Lower (positive) values represent better accuracy of focusing.
Time Frame: 6 week outcome exam
Measure: Least Squares Mean (95% Confidence Interval); unit: Diopters
Arm/Group | Glasses With Hyperopic Lenses | Control
Number analyzed (Participants) | 25 | 23
Diopters | 0.23 [-0.068 to 0.53] | 0.054 [-0.25 to 0.36]

ADVERSE EVENTS:
Arm/Group | Glasses With Hyperopic Lenses | Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/27
Other Adverse Events (participants affected / at risk) | 0/31 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No